CLINICAL TRIAL: NCT03466385
Title: Nasal High Flow Versus Non-Invasive Ventilation in Patients With Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: NHF vs NIV in Patients With Acute Exacerbation of COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Evangelismos Hospital (Other)
Collaborators: Venizeleio General Hospital, Heraklion, Crete (Unknown); Larissa University Hospital (Other); Sotiria General Hospital (Other)
Responsible Party: Principal Investigator, ISCHAKI ELENI, Consultant, ICU Department, Evangelismos Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 48/28-02-2018
Record Dates: First submitted 2018-02-28; First posted 2018-03-15 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Respiratory Failure; Acute Exacerbation Copd
Keywords: Non-invasive ventilation; Nasal High Flow
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasal High Flow (Experimental): Patients randomized to NHF device with initial settings of flow=50-60 L·min-1, temperature=37ο Celsius and FiO2 adjusted to maintain SpO2 between 88%-92%.
  Interventions: Device: Nasal High Flow
- Non-Invasive Ventilation (Active Comparator): Patients randomized to NIV with initial settings EPAP=3cmH2O, IPAP=15cmH2O, I:E=1:2 to 1:3, inspiratory time=0.8-1.2sec and FiO2 adjusted to maintain SpO2 between 88%-92%.
  Interventions: Device: Non-Invasive Ventilation

INTERVENTIONS:
Device: Nasal High Flow — Patients admitted to emergency department with COPD exacerbation combined with mild to moderate acute or acute on chronic hypercapnic respiratory failure will be randomized in one of the two study groups. In case of NHF it will be commence immediately with pre-defined settings
  Arms: Nasal High Flow
Device: Non-Invasive Ventilation — Patients admitted to emergency department with COPD exacerbation combined with mild to moderate acute or acute on chronic hypercapnic respiratory failure will be randomized in one of the two study groups. In case of NIV it will be commence immediately with pre-defined settings
  Arms: Non-Invasive Ventilation

SUMMARY:
Although non-invasive ventilation (NIV) usage has increased significantly over time in COPD exacerbation, a great percentage of patients (~30%) present contraindications to NIV or cannot tolerate it. Nasal high flow (NHF) has been introduced for the management of hypoxemic respiratory failure in adults with favorable effects on ventilation and respiratory mechanics. The above mentioned NHF positive effects has been observed also in stable COPD patients with or without chronic hypercapnia.

In this study, the investigators hypothesize that NHF is not inferior to NIV for respiratory support in patients with COPD exacerbation and acute or acute on chronic hypercapnic respiratory failure.

DETAILED DESCRIPTION:
The use of non-invasive ventilation (NIV) in COPD exacerbation has increased significantly over time since it has been shown to improve acute respiratory acidosis (increases pH and decreases PaCO2), decrease respiratory rate, work of breathing, severity of breathlessness and therefore reduce mortality and intubation rates.

Despite all these favorable effect, a great percentage of patients (~30%) present contraindications to NIV or cannot tolerate it increasing thus the possibility of NIV failure and consequently intubation rates.

Over the past decade, nasal high flow (NHF) oxygen therapy has been introduced for the management of hypoxemic respiratory failure in adults. NHF can generate high flow rates up to 60 L·min-1 and through this mechanism exerts its positive effects on respiratory mechanics, carbon dioxide washout, patient's respiratory rate and work of breathing. Although the above mentioned NHF positive effects has been observed also in stable COPD patients with or without chronic hypercapnia, NHF use in COPD exacerbation is questionable and only a few case reports studies have been published showing favorable effects of NHF on COPD exacerbation.

In this study, the investigators hypothesize that NHF is not inferior to NIV for respiratory support in patients with COPD exacerbation and acute or acute on chronic hypercapnic respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Patient with mild to moderate COPD exacerbation and the following characteristics persisting after initial medical therapy with bronchodilators and controlled oxygen therapy

  * 7,25<pH<7,35
  * PaCO2>45mmHg
  * RR>23
* Ability to obtain written informed consent by the patient or patient's next of kin

Exclusion Criteria:

* severe facial deformity
* Facial burns
* Fixed upper airway obstruction
* Criteria for imminent intubation and invasive mechanical ventilation (any of the following)

  * respiratory or cardiac arrest
  * gasping respiration
  * pH <7.15
  * depressed consciousness (Glasgow Coma Score <8)
  * psychomotor agitation inadequately controlled by sedation
  * massive aspiration
  * persistent inability to remove respiratory secretions
  * heart rate < 50 ·min-1 with loss of alertness
  * severe hemodynamic instability without response to fluids and vasoactive drugs
  * severe ventricular arrhythmias

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Estimated)
Dates: Start 2018-04-15 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of treatment failure | The first assessment will be held at 2 hours
  As treatment failure is defined any need to switch to other treatment group because of discomfort, intolerance or failure to improve physiologic parameters (especially respiratory rate and ABG) despite optimum settings

SECONDARY OUTCOMES:
Changes on respiratory rate | They will be assessed on baseline, before NIV or NHF initiation, and on 1, 2, 4, 6, 12, 24, 48 hours and once daily after day 3.
  This secondary outcome includes changes on respiratory rate (breaths per minute)
Changes on arterial partial pressure of oxygen | They will be assessed on baseline, before NIV or NHF initiation, and on 1, 2, 4, 6, 12, 24, 48 hours and once daily after day 3.
  This secondary outcome includes changes on arterial partial pressure of oxygen values (unit of measure will be mmHg)
Changes on arterial partial pressure of carbon dioxide | They will be assessed on baseline, before NIV or NHF initiation, and on 1, 2, 4, 6, 12, 24, 48 hours and once daily after day 3.
  This secondary outcome includes changes on arterial partial pressure of carbon dioxide (unit of measure will be mmHg)
Changes on arterial pH | They will be assessed on baseline, before NIV or NHF initiation, and on 1, 2, 4, 6, 12, 24, 48 hours and once daily after day 3.
  This secondary outcome includes changes on arterial pH values
Changes on respiratory accessory muscle use | They will be assessed on baseline, before NIV or NHF initiation, and on 1, 2, 4, 6, 12, 24, 48 hours and once daily after day 3.
  This secondary outcome includes recording of respiratory accessory muscle use (recording will be yes or no)
Patient's dyspnea | They will be assessed on baseline, before NIV or NHF initiation, and on 1, 2, 4, 6, 12, 24, 48 hours and once daily after day 3 (in those subjects whose neurological status allowed them to complete the evaluation)
  Dyspnea will be assessed with a 10-point visual analog scale and also Borg scale for dyspnea
Pulmonary complications | They will be assessed on baseline, before NIV or NHF initiation, and on 1, 2, 4, 6, 12, 24, 48 hours and once daily after day 3.
  Any pulmonary complication will be assessed and correlated with the allocated treatment
Extrapulmonary complications | They will be assessed on baseline, before NIV or NHF initiation, and on 1, 2, 4, 6, 12, 24, 48 hours and once daily after day 3
  Any extrapulmonary complication will be assessed and correlated with the allocated treatment

CONTACTS AND LOCATIONS:
Overall Officials: Spyros Zakynthinos, MD, PhD, FCCP, Principal Investigator — Evangelismos Hospital
Locations (3):
- Greece (3):
  - Venizeleio Hospital, Heraklion, Crete
  - Evangelismos Hospital, Athens
  - University General Hospital of Larisa, Larissa

IPD SHARING:
Plan to Share IPD: Yes
Information that are planned to be shared re study protocol, statistical analysis and clinical study report. They will be shared after 3 months of study publication to anyone who is interested in writing a meta-analysis or review
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 3 months after publication
Access Criteria: To anyone who is interested in writing a meta-analysis or review

REFERENCES:
- [Result] Davidson AC, Banham S, Elliott M, Kennedy D, Gelder C, Glossop A, Church AC, Creagh-Brown B, Dodd JW, Felton T, Foex B, Mansfield L, McDonnell L, Parker R, Patterson CM, Sovani M, Thomas L; BTS Standards of Care Committee Member, British Thoracic Society/Intensive Care Society Acute Hypercapnic Respiratory Failure Guideline Development Group, On behalf of the British Thoracic Society Standards of Care Committee. BTS/ICS guideline for the ventilatory management of acute hypercapnic respiratory failure in adults. Thorax. 2016 Apr;71 Suppl 2:ii1-35. doi: 10.1136/thoraxjnl-2015-208209. No abstract available. PMID 26976648
- [Result] Ischaki E, Pantazopoulos I, Zakynthinos S. Nasal high flow therapy: a novel treatment rather than a more expensive oxygen device. Eur Respir Rev. 2017 Aug 9;26(145):170028. doi: 10.1183/16000617.0028-2017. Print 2017 Sep 30. PMID 28794144
- [Result] Mauri T, Turrini C, Eronia N, Grasselli G, Volta CA, Bellani G, Pesenti A. Physiologic Effects of High-Flow Nasal Cannula in Acute Hypoxemic Respiratory Failure. Am J Respir Crit Care Med. 2017 May 1;195(9):1207-1215. doi: 10.1164/rccm.201605-0916OC. PMID 27997805
- [Result] Fricke K, Tatkov S, Domanski U, Franke KJ, Nilius G, Schneider H. Nasal high flow reduces hypercapnia by clearance of anatomical dead space in a COPD patient. Respir Med Case Rep. 2016 Aug 26;19:115-7. doi: 10.1016/j.rmcr.2016.08.010. eCollection 2016. PMID 27668173
- [Result] Biselli PJ, Kirkness JP, Grote L, Fricke K, Schwartz AR, Smith P, Schneider H. Nasal high-flow therapy reduces work of breathing compared with oxygen during sleep in COPD and smoking controls: a prospective observational study. J Appl Physiol (1985). 2017 Jan 1;122(1):82-88. doi: 10.1152/japplphysiol.00279.2016. Epub 2016 Nov 4. PMID 27815367
- [Result] Braunlich J, Seyfarth HJ, Wirtz H. Nasal High-flow versus non-invasive ventilation in stable hypercapnic COPD: a preliminary report. Multidiscip Respir Med. 2015 Sep 3;10(1):27. doi: 10.1186/s40248-015-0019-y. eCollection 2015. PMID 26339486
- [Result] Fraser JF, Spooner AJ, Dunster KR, Anstey CM, Corley A. Nasal high flow oxygen therapy in patients with COPD reduces respiratory rate and tissue carbon dioxide while increasing tidal and end-expiratory lung volumes: a randomised crossover trial. Thorax. 2016 Aug;71(8):759-61. doi: 10.1136/thoraxjnl-2015-207962. Epub 2016 Mar 25. PMID 27015801
- [Result] Pisani L, Fasano L, Corcione N, Comellini V, Musti MA, Brandao M, Bottone D, Calderini E, Navalesi P, Nava S. Change in pulmonary mechanics and the effect on breathing pattern of high flow oxygen therapy in stable hypercapnic COPD. Thorax. 2017 Apr;72(4):373-375. doi: 10.1136/thoraxjnl-2016-209673. Epub 2017 Jan 19. PMID 28104830
- [Result] Lepere V, Messika J, La Combe B, Ricard JD. High-flow nasal cannula oxygen supply as treatment in hypercapnic respiratory failure. Am J Emerg Med. 2016 Sep;34(9):1914.e1-2. doi: 10.1016/j.ajem.2016.02.020. Epub 2016 Feb 12. No abstract available. PMID 26947372
- [Derived] Pantazopoulos I, Boutlas S, Mavrovounis G, Papalampidou A, Papagiannakis N, Kontou M, Bibaki E, Athanasiou N, Meletis G, Gourgoulianis K, Zakynthinos S, Ischaki E. Nasal high flow or noninvasive ventilation? navigating hypercapnic COPD exacerbation treatment: A randomized noninferiority clinical trial. Respir Med. 2024 Oct;232:107762. doi: 10.1016/j.rmed.2024.107762. Epub 2024 Aug 5. PMID 39111544